CLINICAL TRIAL: NCT03997487
Title: Developing and Evaluating Trachoma Diagnosis Training Tools in Preparation for the Trachoma Elimination Endgame: Development of a Smartphone Application to Capture Quality Images of Everted Eye Lids and Assessment of Its Acceptability and Feasibility
Brief Title: Smartphone App for Taking Images of Conjunctivae
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: National Institute for Medical Research, Tanzania (Other Government); Federal Minstry of Health of Ethiopia (Other Government); Jos University Teaching Hospital (Other); University College London Hospitals (Other); RTI International (Other); Sightsavers (Unknown); World Health Organization (Other); Pan American Health Organization (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2019-KEP-284 - 2
Record Dates: First submitted 2019-06-19; First posted 2019-06-25 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-05

CONDITIONS: Trachoma
MeSH Terms: conditions — Trachoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children examined (Experimental): All children examined for clinical signs of trachoma will be invited to participate to have photos of conjunctivae taken with the TOFTEE smartphone app and a DSLR camera.
  Interventions: Other: TOFTEE

INTERVENTIONS:
Other: TOFTEE — Smartphone app for taking quality images of conjunctivae

SUMMARY:
Trachomatous inflammation-follicular (TF) is diagnosed by looking for clinical signs of infection of everted eyelids (conjunctivae) of children.

The overall objective of this project is to develop a smartphone application and assess its acceptability and feasibility.

Fieldwork will take place during routine Tropical Data trainings and population-based prevalence surveys supported by Tropical Data.

Healthy adult volunteers in London will have photos of their conjunctivae taken to develop the app initially, with iterative improvements to the app based on image quality achieved. For fieldwork, images of the conjunctivae of children will be have photos of their conjunctivae taken with a digital single lens reflex (DSLR) camera and the newly developed smartphone app. Grading of the photos will be compared with field grading, to compare grading agreement, to assess utility for supervision, quality assurance and training purposes.

DETAILED DESCRIPTION:
The investigators want to see whether it would be possible to take photos using Android smartphones, routinely used in trachoma surveys for collecting data, for quality assurance, supervision and training purposes. The investigators will develop an app in the United Kingdom (UK) by taking photos of the conjunctivae of healthy adult volunteers to iteratively improve the quality of images based on the image metadata and review by trachoma experts. The app will then be field tested, and trachoma grading based on the app photos, DSLR photos, and clinical grading, compared. Any management (treatment) will be based on routine clinical diagnosis only - the images are for research purposes only. The investigators will also ask participants for their views on acceptability of having photos of conjunctivae taken with the phone, and conduct a cost-consequences analysis of potential implementation of the app in routine trachoma surveys.

Objectives and approach:

2.1 To develop a mobile phone application to capture images of everted eyelids (conjunctivae) of children being examined as part of the Tropical Data field inter-grader agreement (IGA) test, or sampled as part of trachoma prevalence surveys.

2.2 To evaluate the quality of the mobile phone application images compared with field grading and DSLR images.

2.3 To assess the acceptability and feasibility of a mobile phone application for photographing everted eyelids (conjunctivae) from children being examined as part of the Tropical Data IGA test, or sampled as part of trachoma prevalence surveys.

2.4 To conduct a cost-consequences analysis of setting up an infrastructure for capturing and transmitting images in order to make the system economically viable.

ELIGIBILITY:
Inclusion Criteria:

Objectives 2.1 and 2.2:

* For the London-based app development, any eligible healthy adult who provides written informed consent will be eligible.
* For the field-based app development, any child aged 1-9 years being examined as part of the Tropical Data IGA test, or sampled as part of trachoma prevalence surveys, and for whom written informed consent has been provided by a guardian, will be eligible.

Objective 2.3:

* All Tropical Data trainers and trainees attending the Tropical Data (initial and refresher) training events and who provide written informed consent, will be eligible.
* Community leaders and children's guardians who provide written informed consent will be eligible.

Exclusion Criteria:

* For each of the objectives, if the inclusion criteria are not fulfilled, the participant will not be eligible to participate.

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2019-07-12 (Actual); Study Completion 2019-07-12 (Actual)

PRIMARY OUTCOMES:
TOols For Trachoma Elimination Endgame (TOFTEE) app image quality | 30 minutes
  Photo quality will be assessed by trachoma grading experts. The technical parameters such as lighting, resolution, focus, etc. will be assessed using objective software or extracted from the photograph metadata.
Kappa score of TOFTEE image compared with field grading | 5 minutes
  Concordance in diagnosis of trachoma between field grading and app image
Kappa score of TOFTEE image compared with DSLR grading | 5 minutes
  Concordance in diagnosis of trachoma between app image and DSLR image
Kappa score of DSLR image compared with field grading | 5 minutes
  Concordance in diagnosis of trachoma between field grading and DSLR image

SECONDARY OUTCOMES:
Association (reported as proportions, unadjusted and adjusted odds ratios) between child characteristics and TOFTEE image quality | 15 minutes
  Association (reported as proportions, unadjusted and adjusted odds ratios) between child characteristics acceptable photo quality
Acceptability and feasibility of TOFTEE app in communities | 45 minutes
  Common themes, as determined through thematic analysis of focus group discussion transcripts, relating to acceptability and feasibility of TOFTEE app in communities
Acceptability and feasibility of TOFTEE app in Tropical Data system | 45 minutes
  Common themes, as determined through thematic analysis of focus group discussion transcripts, relating to acceptability and feasibility of TOFTEE app as part of the Tropical Data system
Cost of TOFTEE app implementation | 5 days
  Cost (overall and broken down by category: personnel; supplies; transit; telecommunications) of TOFTEE app implementation into the Tropical Data system

CONTACTS AND LOCATIONS:
Overall Officials: Emma Harding-Esch, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Arusha region, Arusha, Tanzania

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data will be shared with relevant study team members for the purposes of data analysis. Data Transfer Agreements will be completed, where appropriate.
Supporting Information: Study Protocol
Time Frame: Data will be shared with team members as they are collected.
Access Criteria: Data access requests from outside the study team for the specified data analyses will be reviewed by the Principal Investigator. Requestors will be required to sign a Data Access Agreement.